CLINICAL TRIAL: NCT01059513
Title: Hypo-fractionated Stereotactic Body Radiotherapy for Localized Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 10-001787
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-05

CONDITIONS: Prostate Cancer
Keywords: T1c; T2a; T2b
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an observational study in which a questionnaire is used to obtain quality of life data after patients undergo a hypo-fractionated course of stereotactic body radiotherapy (SBRT) for the treatment of their prostate cancer. The SBRT itself is considered standard of care for these patients and as such, is not an official component of the study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will have clinical stage T1c, T2a, or T2b, a pre-biopsy PSA level <10 ng/mL and a biopsy Gleason score of 3+3 (or 3+4 if fewer than 30% of biopsy cores are involved).
* The ability to understand and willingness to sign a written informed consent are necessary.

Exclusion Criteria:

* Patients with tumor parameters that fall outside of the inclusion criteria.
* Patients with evidence on imagining (bone scan, CT, or MRI) suggestive of disseminated disease.
* Patients who have had any form of prior prostate treatment (surgery, radiotherapy, cryotherapy, high intensity focused ultrasound, TURP).
* A prior course of hormone therapy (androgen deprivation) of greater than 3 months duration.
* The use of other concurrent investigational agents.
* There are no exclusions due to co-morbid disease or illnesses except for patients with severe inflammatory bowel disease.
* No life expectancy restrictions will apply.
* Performance status will not be considered.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will have clinical stage T1c, T2a, or T2b, a pre-biopsy PSA level <10 ng/mL and a biopsy Gleason score of 3+3 (or 3+4 if fewer than 30% of biopsy cores are involved).
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2010-01-26 (Actual); Primary Completion 2020-03-19 (Actual); Study Completion 2020-03-19 (Actual)

PRIMARY OUTCOMES:
To quantify patient quality of life after prostate SBRT using validated questionnaire tools | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher King, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California, United States